CLINICAL TRIAL: NCT00545389
Title: A Phase II, Randomized, Multi-centre, Double-blind, Parallel-group, Dose-ranging, Exploratory Study in Subjects With Mild to Moderate Ulcerative Colitis Treated With SPD476 (Mesalazine) Once Daily
Brief Title: Phase II Dose-Ranging Study in Subjects With Mild to Moderate Ulcerative Colitis Treated With SPD476
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD476-202
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: SPD476 is a polymeric matrix formulation that displays both delayed- and extended-release of mesalazine
  Other Names: LIALDA

SUMMARY:
Evaluate the percentage of subjects in remission at the end of an 8-week treatment period for three dose groups (SPD476 1.2 g/day, 2.4 g/day or 4.8 g/day, administered once daily).

ELIGIBILITY:
Inclusion Criteria:

* male & female subjects greater than or equal to 18 years of age with newly diagnosed or relapsing mild to moderate ulcerative colitis
* general medical assessment satisfactory and no clinically significant and relevant abnormalities

Exclusion Criteria:

* severe ulcerative colitis
* subject in relapse for > 6 weeks
* use of systemic or rectal steroids within last 4 weeks prior to baseline
* subjects with proctitis, previous colonic surgery, Crohn's disease, bleeding disorders, active ulcer disease
* subjects hypersensitive to salicylates/aspirin
* subjects with moderate or severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-02-10 (Actual); Primary Completion 2004-10-20 (Actual); Study Completion 2004-10-20 (Actual)

PRIMARY OUTCOMES:
% of subjects in remission (UC-DAI score) | Week 8

SECONDARY OUTCOMES:
Change in UC-DAI score by dose and by diagnosis, change in symptoms, change in sigmoidoscopic (mucosal) appearance, change in histology | 8 weeks
Plasma levels & mucosal levels of 5-ASA and Ac-5-ASA | 8 weeks
Safety and tolerability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Imelda General Hospital, Bonheiden, Belgium

REFERENCES:
- [Result] D'Haens G, Hommes D, Engels L, Baert F, van der Waaij L, Connor P, Ramage J, Dewit O, Palmen M, Stephenson D, Joseph R. Once daily MMX mesalazine for the treatment of mild-to-moderate ulcerative colitis: a phase II, dose-ranging study. Aliment Pharmacol Ther. 2006 Oct 1;24(7):1087-97. doi: 10.1111/j.1365-2036.2006.03082.x. PMID 16984503
- See also: FDA-approved label, US only — http://www.lialda.com/
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html